CLINICAL TRIAL: NCT06069297
Title: Multimodal Prehabilitation in Localized Pancreatic Cancer Patients Undergoing Surgery: a Randomized Controlled Trial
Brief Title: Prehabilitation in Pancreatic Surgery
Acronym: PIPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Nicolò Pecorelli, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GR-2021-12374985
Record Dates: First submitted 2023-08-25; First posted 2023-10-05 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer; Periampullary Cancer; Frailty Syndrome; Malnutrition; Perioperative/Postoperative Complications
Keywords: Prehabilitation; Physical function; Nutritional status; Functional capacity; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Frailty; Malnutrition; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomized (ratio 1:1) and allocated either to the intervention group (Multimodal Prehabilitation) or to the usual care group
Who Masked: Outcomes Assessor
Masking Description: The trial is designed as a randomized, controlled, assessor-blind trial.
  Patient and investigator blinding will not be feasible due to the nature of the intervention and the direct involvement of the prehabilitation team. However, to minimize potential blinding and performance biases, enrolled patients will be informed that we will compare two types of strategies (prehabilitation and usual care), both aiming at improving their health conditions and fitness before surgery, and neither will be presented as potentially superior.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal Prehabilitation (Experimental): The intervention consists of a supervised multimodal prehabilitation program (exercise, nutritional support, and psychosocial counseling) conducted for a minimum of four weeks prior to surgery, during the waiting time following patient enrolment.
  Interventions: Other: Multimodal Prehabilitation
- Usual care (No Intervention): Usual preoperative care. Patients in the control group will be treated according to usual care and will be given informative material regarding a healthy lifestyle and how to best prepare for surgery.

INTERVENTIONS:
Other: Multimodal Prehabilitation — Preoperative multimodal intervention including exercise training, nutritional therapy and psychosocial counseling, aimed at preventing or attenuating surgery-driven functional decline. A personalized intervention program will be prescribed based on specific physical, nutritional and psychological conditions recognized during the multimodal assessment. Patients will follow a 2 to 3-day per week exercise program for 4-6 weeks including endurance, resistance, and inspiratory muscle training, tailored to individual preferences and clinical conditions. Based on dietary habits and nutritional status, a certified nutritionist will provide a comprehensive diet management program. A food-based intervention with a balanced macronutrient composition coupled with oral nutritional supplements will be prescribed to achieve the estimated daily energy and protein requirements. Patients will meet with a psychologist to explore their emotional and psychosocial needs related to their current situation.
  Arms: Multimodal Prehabilitation

SUMMARY:
In patients with pancreatic cancer, older age, multiple comorbidities, frailty, malnutrition and poor functional status are common, especially in individuals receiving neoadjuvant chemotherapy. These characteristics represent potentially modifiable risk factors for poor postoperative outcomes.

The goal of this clinical randomized controlled trial is to evaluate the extent to which a four-week multimodal prehabilitation program impacts on postoperative morbidity, functional and nutritional status and health-related quality of life in patients with localized pancreatic or periampullary cancer scheduled for curative surgery.

In addition, the impact of prehabilitation on circulating sarcopenia and cancer cachexia biomarkers in PDAC patients will be explored.

Included patients will be randomized (ratio 1:1) and allocated either to the intervention group (Multimodal Prehabilitation), which will receive prehabilitation, or to the control group, which will receive no prehabilitation.

DETAILED DESCRIPTION:
BACKGROUND:

Pancreatic ductal adenocarcinoma (PDAC) is a highly lethal cancer, with 5-year survival around 10%. The combination of surgical resection and chemotherapy represents the most efficacious therapy to improve prognosis for localized PDAC. Patients with pancreatic cancer are generally older adults in whom frailty, sarcopenia and/or malnutrition are common. These features have all been associated with poor postoperative complications and reduced survival. Therefore, the preoperative period and the time window after the end of chemotherapy constitute a unique opportunity to condition modifiable risk factors, improve functional capacity and address deficiencies in physiologic reserves, which might otherwise preclude surgery or significantly impede recovery.

Prehabilitation is defined as the process of enhancing patients' functional capacity to enable them to withstand a stressful event. Multimodal prehabilitation, which defines a program including physical, nutritional, and psychological interventions, has shown the most promising results in gastrointestinal cancer surgery. However, no high-quality evidence is currently available for PDAC patients.

STUDY OBJECTIVES:

Primary Aim: to evaluate if a 4-week multimodal structured prehabilitation program including physical exercise, nutritional and psychological interventions will result in a clinically significant increase in functional capacity, nutritional status and patient-reported health-related quality of life before surgery when compared to a usual care control group, and evaluate the extent to which multimodal prehabilitation impacts on postoperative morbidity and patient recovery compared to usual care.

Secondary Aim: to analyze whether multimodal prehabilitation may impact on the concentration and activity of a panel of specific circulating molecules involved in cancer cachexia and skeletal muscle wasting, chronic inflammation.

STUDY DESIGN:

A randomized controlled trial will be performed in PDAC and periampullary cancer patients with indication to upfront pancreatic resection or pancreatic resection after completion of neoadjuvant chemotherapy.

Included patients will be randomized (ratio 1:1) and allocated either to the intervention group (Multimodal Prehabilitation), which will receive prehabilitation, or to the control group, which will receive no prehabilitation. All patients will receive the same intraoperative and postoperative care based on an established enhanced recovery pathway.

Inclusion and exclusion criteria as stated in the eligibility section will be assessed and patients consented to participate in the study if they fulfill inclusion criteria.

RANDOMIZATION AND BLINDING:

The trial is designed as a randomized, controlled, assessor-blind trial. Participants will be randomly assigned to either multimodal prehabilitation or no prehabilitation group with a 1:1 allocation using permuted blocks of random sizes. Randomization will be stratified by neoadjuvant chemotherapy and tumor location (periampullary or pancreatic head-neck cancer versus pancreatic body-tail cancer). Allocation concealment will be ensured as the randomization code will not be released until the patient has been recruited into the trial, which takes place after all baseline measurements have been completed and informed consent has been signed.

PREOPERATIVE ASSESSMENT:

All patients will be evaluated at baseline (T0) by:

* Patient medical history including comorbidities, presence of signs or symptoms, and frailty assessment using Fried's criteria.
* Physical performance tests including functional walking capacity (six-minute walk test), timed up and go test, gait speed assessment and handgrip strength test.
* Assessment of nutritional status by nutrition history, measurement of anthropometric parameters, completion of nutritional screening questionnaires (MNA, PG-SGA), and standard biochemical markers of malnutrition and inflammation including albumin, prealbumin, total lymphocyte count, and C-reactive protein.
* Body composition measurements assessed using two methods:

  * multi-frequency bioelectrical impedance analysis (BIA) providing data on extracellular and intracellular water as % of total body water, fat mass (FM) as % of body weight, skeletal muscle mass (SK) as % of fat-free mass (FFM) and phase angle (PA°), intramuscular fat mass (IMAT), basal metabolic rate (BMR) energy expenditure and hypotalamic- pituitary- adrenal axis index (HPA);
  * CT scan image analysis (using preoperative cancer staging and restaging chest and abdomen CT scans) performing automated imaging segmentation using Data Analysis Facilitation Suite (DAFS) by Voronoi Health Analytics, Inc. (https://www.voronoihealthanalytics.com/).
* Overall activity of the autonomic nervous system and heart rate variability through photoplethysmography (PPG) stress flow test. This exam allows the study and direct monitoring of all functions of the autonomic nervous system and the related process of biofeedback.
* Patient reported outcome questionnaires to measure health related quality of life and patient engagement. The following questionnaires will be administered

  * Patient reported outcome measurement information system (PROMIS)29+2, a validated questionnaire designed to measure self-reported physical, mental and social health and wellbeing.
  * Duke activity status index (DASI), a brief questionnaire designed to assess physical function by answering whether they are able to perform 12 listed activities of various intensity (i.e., ambulation, household tasks and leisure activities).
  * EORTC QLQ C30, a generic core questionnaire that measures health-related quality of life in patients with any cancer.
  * EORTC QLQ PAN-26, the pancreatic cancer module that supplements the EORTC QLQ-C30.
  * - Medically unexplained symptoms (MUS) questionnaire investigates the presence of vague symptoms to describe a cluster of manifestations such us chronic fatigue, sleep or appetite disorders, irritable bowel or constipation, tone or mood disorders, non-specific pain syndromes which are sometimes underestimated.
  * Patient activation measures (PAM)-13, a 13-item questionnaire measuring patients' self-reported knowledge, motivation, and skills for self-management.
  * Hospital Anxiety and Depression Scale (HADS) questionnaire to measure anxiety and depression.
* Blood sample analysis of circulating cytokines, chemokines, interferons, colony stimulating factors, main hormones involved in metabolic homeostasis and cancer cachexia.

Four weeks after baseline assessment, on the day before surgery (T1), all patients will repeat all evaluations previously performed at T0.

STUDY INTERVENTION Included patients will be randomized (ratio 1:1) and allocated either to the intervention group (Multimodal Prehabilitation), which will receive prehabilitation, or to the control group, which will receive no prehabilitation. Patients in the control group will be treated according to usual standard of care and will be given informative material regarding healthy lifestyle and how to best prepare for surgery.

The intervention will consist of a multimodal prehabilitation, a 4-week long preoperative intervention including exercise training, nutritional therapy and anxiety reducing techniques, aimed at preventing or attenuating surgery-driven functional decline as described in the arms and intervention section.

VISITS AND FOLLOW-UP:

Throughout patient hospital stay, postoperative outcomes including complications, will be recorded. After discharge, patients will be followed-up as routine care by phone calls from a nurse navigator.

At 30 days (T2), 60 (T3) and 90 days (T4) after surgery, patient recovery will be re-evaluated during scheduled outpatient visits. Patients will be assessed for:

* Functional capacity by the 6MWT and other physical performance tests including TUG, gait speed assessment and handgrip strength test.
* Nutritional status by measurement of anthropometric parameters including body weight (kg), height (cm), and body mass index (kg/m2)
* Body composition by multi-frequency bioelectrical impedance vector analysis (BIVA)
* Health related quality of life through patient reported outcome questionnaires

STATISTICAL METHODS:

Continuous variables will be summarized using either median and interquartile range (IQR) or mean ± standard deviation (SD), depending on data distribution. Categorical variables will be reported as frequencies and percentages. All analyses will follow the intention-to-treat principle.

The between-group difference in the primary outcome will be assessed using a linear regression model after applying a log(+1) transformation to the 90-day Comprehensive Complication Index (CCI®️), adjusting for relevant confounders. Continuous secondary outcomes will be analyzed using appropriate generalized linear models, while binary outcomes will be evaluated using logistic regression to estimate odds ratios (ORs) with 95% confidence intervals (CIs).

To account for the repeated measures design, linear mixed-effects models will be employed, incorporating treatment group and time as fixed effects, and patient ID as a random effect. This model will estimate the mean differences in outcomes over time between groups. The effect of the intervention will be reported as adjusted least square mean differences along with corresponding 95% CIs.

To minimize attrition bias, missing data will be handled using multiple imputation with chained equations and predictive mean matching. A sensitivity analysis will be conducted to assess the impact of missing data on the primary outcome. A per-protocol analysis will also be performed, including only patients who completed at least 80% of the prehabilitation sessions and excluding those lost to follow-up or who withdrew.

A pre-specified subgroup analysis will explore whether the effect of prehabilitation versus standard care on the primary outcome and functional capacity differs across the following patient subgroups:

* Frail versus non-frail, defined by Fried Frailty Score Index (FFSI ≥ 2 vs < 2);
* Neoadjuvant therapy versus upfront surgery;
* Proximal versus distal pancreatectomy;
* Elderly versus younger patients, defined as > 75 years vs ≤ 75 years;
* Low versus high baseline functional capacity, based on 6-minute walk distance (6MWD < 400 m vs ≥ 400 m) or Duke Activity Status Index (DASI < 34 vs ≥ 34);
* High versus low psychological distress, defined by HADS subscale scores (≥ 8 vs < 8);
* Nutritional status, defined by PG-SGA scores (< 4 well-nourished, 4-8 moderately malnourished, > 8 severely malnourished);
* Sarcopenic versus non-sarcopenic, defined by BIVA-derived ASMMI values (< 7.0 kg/m² in men and < 5.7 kg/m² in women) and CT scan-derived skeletal muscle areas.
* Overweight versus non-overweight patients, defined by BMI values (>24.99 kg/m²)

Patient satisfaction will be described using means and SDs for continuous variables (or medians and IQRs for skewed distributions) and frequencies and percentages for categorical data. Barriers to adherence among participants who did not meet the 80% session completion threshold will be explored through qualitative interviews, transcribed and categorized according to the COM-B model (Capability, Opportunity, Motivation).

Statistical significance will be set at a p-value < 0.05. All analyses will be conducted using STATA® version 18 (StataCorp, College Station, TX, USA).

SAMPLE SIZE:

The size of the sample was calculated on the basis of the primary aim of the study: the reduction of postoperative complications as determined with the CCI score at 90 days after surgery. In our preliminary data on PDAC surgical population, the mean (SD) CCI is 21.0 (SD 16), and the target reduction is 30%. An alpha of 0.05 and power of 0.80 (two-sided test) was used. Accounting for a 15% of dropout rate, the required sample size was 238 patients, 119 for each arm.

ECONOMIC EVALUATIONS:

Hospital-related costs will be collected for all patients included in the study over a 90-day postoperative period. These costs include expenses directly associated with patient care, such as the prehabilitation program (staff time, facilities, equipment, and sessions), surgical procedures, length of hospital stay, management of complications, remissions, and follow-up visits within 90 days after surgery. Comparing hospital costs between patients receiving prehabilitation and those undergoing standard care will provide valuable insight into the economic impact of prehabilitation on healthcare resource utilization during the early postoperative period.

A cost-utility analysis will be conducted to evaluate the economic value of the prehabilitation program compared to standard care over the 90-day postoperative period. Health-related quality of life (HRQoL) will be assessed using the PROMIS-29+2, which provides the PROPr (Patient-Reported Outcomes Measurement Information System Preference score), a preference-based utility measure derived from PROMIS item responses. These utility values quantify the quality of health on a scale where 0 represents death and 1 represents perfect health. By combining these utility scores with the length of the follow-up period, quality-adjusted life years (QALYs) can be estimated, reflecting both the quantity and quality of life experienced by each patient during this timeframe. This approach allows for capturing the changes in patients' health status due to the intervention or standard care. Hospital costs incurred during the same 90-day period, including all healthcare resource use such as hospital stay, procedures, complications management, and prehabilitation costs, will be integrated into the analysis. The incremental cost-effectiveness ratio (ICER) will then be calculated by dividing the difference in average costs between the two groups by the difference in average QALYs gained. The ICER represents the additional cost required to gain one additional quality-adjusted life year through prehabilitation compared to standard care, providing a summary measure of the intervention's cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication for curative resection for pancreatic or periampullary cancer
* Signed Informed consent

Exclusion Criteria:

* Metastatic or unresectable disease found preoperatively
* Comorbidities contraindicating prehabilitation regimen (exercise and nutritional intervention) such as orthopedic, cognitive disabilities, chronic renal failure (dialysis or creatinine >250 mmol)
* ASA score 4-5
* Pregnancy
* Illiteracy (inability to read and understand Italian language)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index (CCI) | 90 days after surgery
  Postoperative complications occurring during the index admission or in a subsequent readmission, when related to surgery, will be recorded up to 90 days after surgery and graded by severity using the Dindo-Clavien classification and the Comprehensive Complication index (CCI).
  The Dindo-Clavien system grades complications according to the therapy needed for treatment: Grade I, are complications that require bedside management; Grade II, are complications that require pharmacologic treatment; Grade III, are complications that require surgical or radiologic intervention and; Grade IV, are complications that require intensive care treatment. Dindo-Clavien Grade III or above are considered severe postoperative complications.
  The CCI, derived from the Dindo-Clavien system, is a validated metric summarizing the complete spectrum of complications that occurred and their severity in a single score ranging from 0 to 100.

SECONDARY OUTCOMES:
Time to patient functional recovery (TFR) | 90 days after surgery
  TFR will be measured by subtracting the date of surgery from the date when participants achieve standardized criteria (tolerance of oral intake, recovery of lower gastrointestinal function, adequate pain control on oral analgesia, ability to mobilize and self-care and no evidence of untreated medical problems)
Lenght of stay (LOS) | 90 days after surgery
  LOS will be measured by subtracting the date of surgery from the date of discharge
Functional capacity | One day before surgery; 30 days after surgery; 60 days after surgery; 90 days after surgery
  Functional capacity will be measured by the 6-minute walking test, timed up and go test (TUG), gait speed assessment, handgrip strength test, and compared between groups on the day before surgery, at 30-60-90 days after surgery.
Nutritional status | One day before surgery; 30 days after surgery; 60 days after surgery; 90 days after surgery.
  Nutritional status will be measured by weight (kg), height (cm), and body mass index (kg/m2), and nutritional screening questionnaires (mini nutritional assessment - MNA, patient-generated - subjective global assessment - PG-SGA) and compared between groups at baseline, on the day before surgery, at 30, 60, 90 days after surgery..
Bioimpedance analysis (BIA) derived body composition | One day before surgery; 30 days after surgery; 60 days after surgery; 90 days after surgery
  Extracellular and intracellular water as % of total body water, fat mass (FM) as % of body weight, skeletal muscle mass (SK) as % of fat-free mass (FFM), phase angle (PA°) and intramuscular fat mass (IMAT) will be assessed using bioimpedance analysis and compared between groups at baseline, on the day before surgery, at 30, 60, 90 days after surgery.
Computed tomography derived body composition | One day before surgery.
  Skeletal muscle area (cm2), visceral fat area (cm2) and intra-muscular fat infiltration will be measured at the level of the third lumbar vertebra using preoperative CT scan imaging and compared between groups at baseline and on the day before surgery.
Generic health-related quality of life | One day before surgery; 30 days after surgery; 60 days after surgery; 90 days after surgery
  Generic health-related quality of life will be measured using the Patient Reported Outcome Measure Information System (PROMIS)-29+2 Profile v2.1 (PROPr), a questionnaire designed to measure self-reported physical, mental and social health and wellbeing. Questions are ranked on a 5-point Likert Scale. Each domain (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities) is scored from 4 to 20. For negative domains (i.e. Depression), lower scores represent better outcomes, higher scores represent worse outcomes. For positive domains (i.e. Physical function), lower scores represent worse outcomes, higher scores represent better outcomes.
Disease-specific health-related quality of life | One day before surgery; 30 days after surgery; 60 days after surgery; 90 days after surgery
  Disease-specific health-related quality of life will be measured using the EORTC QLQ C30 and PAN-26 questionnaires, which have been validated to assess quality of life in cancer patients.
  EORTC QLQ C30 is a generic core questionnaire that measures health-related quality of life in patients with any cancer. It comprises a total of 30 items on 15 quality of life scales. EORTC QLQ PAN-26, is the pancreatic cancer module that supplements the EORTC QLQ-C30. The module comprises 26 questions that share the 4-level ordinal response options with QLQ-C30.
Patient reported anxiety and depression | One day before surgery; 30 days after surgery; 60 days after surgery; 90 days after surgery.
  Patient reported anxiety and depression will be measured using the Hospital Anxiety and Depression Scale (HADS) questionnaire and compared at baseline, preoperatively, at 30, 60, 90 days after surgery.
  It comprises seven questions for anxiety and seven questions for depression, and the two domains are scored separately. It has been validated in many languages, countries, and settings.
Patient engagement and activation | One day before surgery; 30 days after surgery; 60 days after surgery; 90 days after surgery.
  Patient engagement and activation will be measured using the Patient Activation Measure (PAM)-13, a 13-item questionnaire measuring patients' self-reported knowledge, motivation, and skills for self-management. The Italian version of the questionnaire has been validated in a sample of chronically ill patients. The minimal important difference is 5 points.
  PAM-13 will be administered and compared between groups at baseline, preoperatively, 30 days after surgery; 60 days after surgery; 90 days after surgery.
Pro-inflammatory cytokines | One day before surgery
  Circulating levels of tumor necrosis factor alpha (TNF-α), interleukin 1 (IL-1), interleukin 6 (IL-6), interferon gamma (IFN-γ), and macrophage inflammatory protein α (MIP-1α) will be assessed by luminex immunoassays and compared between groups at baseline and one day before surgery.
Cancer cachexia related factors | One day before surgery
  Enzyme-linked immunosorbent assay (ELISA) will be used to measure the serum levels of the following cachexia-related factors: Activin A, carnosine dipeptidase-1 and zinc-α2-glycoprotein. The circulating levels will be compared between groups at baseline and one day before surgery.

OTHER OUTCOMES:
Hospital costs | 90 days after surgery
  Hospital-related costs will be collected for all patients included in the study over a 90-day postoperative period. These costs include expenses directly associated with patient care, such as the prehabilitation program (staff time, facilities, equipment, and sessions), surgical procedures, length of hospital stay, management of complications, remissions, and follow-up visits within 90 days after surgery. Comparing hospital costs between patients receiving prehabilitation and those undergoing standard care will provide valuable insight into the economic impact of prehabilitation on healthcare resource utilization during the early postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Falconi, MD, Study Chair — San Raffaele Hospital
Locations (1):
- San Raffaele Hospital, Milan, Lombardy, Italy

REFERENCES:
- [Background] Mizrahi JD, Surana R, Valle JW, Shroff RT. Pancreatic cancer. Lancet. 2020 Jun 27;395(10242):2008-2020. doi: 10.1016/S0140-6736(20)30974-0. PMID 32593337
- [Background] Lambert JE, Hayes LD, Keegan TJ, Subar DA, Gaffney CJ. The Impact of Prehabilitation on Patient Outcomes in Hepatobiliary, Colorectal, and Upper Gastrointestinal Cancer Surgery: A PRISMA-Accordant Meta-analysis. Ann Surg. 2021 Jul 1;274(1):70-77. doi: 10.1097/SLA.0000000000004527. PMID 33201129
- [Background] Pecorelli N, Guarneri G, Vallorani A, Limongi C, Licinio AW, Di Salvo F, Tamburrino D, Partelli S, Crippa S, Falconi M. Validation of the PROMIS-29 Questionnaire as a Measure of Recovery After Pancreatic Surgery. Ann Surg. 2023 Nov 1;278(5):732-739. doi: 10.1097/SLA.0000000000006020. Epub 2023 Jul 19. PMID 37465965
- [Derived] Pecorelli N, Fermi F, Abati M, Bonomi B, Fossati L, Corti G, Guarneri G, Macchini M, Damascelli A, Palumbo D, Gaviraghi S, Di Mattei V, De Cobelli F, Tettamanti A, Falconi M. Multimodal Prehabilitation In Pancreatic cancer Patients undergoing surgery (PIPS): study protocol for a randomized controlled trial. Trials. 2026 Jan 31. doi: 10.1186/s13063-026-09467-z. Online ahead of print. PMID 41618415